CLINICAL TRIAL: NCT05905757
Title: Intraoperative and Postoperative Effects of Adjuvant Dexmedetomidine and Tramadol in Subcostal Transversus Abdominis Plan Block
Brief Title: Adjuvant Dexmedetomidine and Tramadol in Subcostal Transversus Abdominis Plan Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2023/2
Record Dates: First submitted 2023-05-16; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Transversus Abdominis Plane Block
Keywords: Transversus abdominis plane block; adjuvant; Dexmedetomidine; Tramadol
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Tramadol

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Experimental): Group T (Adjuvant tramadol): Bilateral subcostal TAP block was performed using solutions prepared by adding 0.250% bupivacaine + 40 mL adjuvant 1.5mg/kg (maximum 100 mg) tramadol.
  Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), HR, SpO2 values were recorded.
  Demographic data of the patients [age, weight, height, body mass index (BMI), smoking use] and operation times were recorded.
  All patients were administered 1000 mg parol IV as standard analgesic before extubation.
  The patients were followed up for side effects (such as nausea-vomiting, chills, itching and desaturation) including drug allergies.The patients were evaluated at 0, 3 and 6 hours after the operation with a 0-10 verbal rating scale visual analog scale (VAS) and the data were recorded. In all groups, VAS˃ 4 value was evaluated in favor of analgesic need and 50 mg Dexketoprofen IV bolus was administered in accordance with conventional treatment.
  Interventions: Drug: Tramadol + Bupivacaine
- Group D (Experimental): Group D (adjuvant dexmedetomidine): Bilateral subcostal TAP block was performed using solutions prepared by adding 0.250% bupivacaine + 0.5 mcg/kg and (maximum 50 mcg) dexmedetomidine.
  All patients were administered 1000 mg parol IV as standard analgesic before extubation.
  The patients were followed up for side effects (such as nausea-vomiting, chills, itching and desaturation) including drug allergies.
  The patients were evaluated at 0, 3 and 6 hours after the operation with a 0-10 verbal rating scale visual analog scale (VAS) and the data were recorded. VAS 0-2: no pain, 3-4: mild pain, 5-6: moderate pain, 7-8: severe pain, 9-10: excruciating pain. Additional analgesic requirement in the postoperative period was calculated by measuring VAS>4 values. In all groups, VAS˃ 4 value was evaluated in favor of analgesic need and 50 mg Dexketoprofen IV bolus was administered in accordance with conventional treatment.
  Interventions: Procedure: Dexmedetomidin + bupivacaine

INTERVENTIONS:
Procedure: Dexmedetomidin + bupivacaine — dexmedetomidine was added as adjuvant to bupivacaine in transversus abdominis plane block (TAP)
  Arms: Group D
Drug: Tramadol + Bupivacaine — tramadol was added as adjuvant to bupivacaine in transversus abdominis plane block (TAP)
  Arms: Group T

SUMMARY:
In this study, dexmedetomidine and tramadol were added as adjuvant to bupivacaine in transversus abdominis plane block (TAP), intraoperative hemodynamics, opioid consumption, muscle relaxant use, postoperative analgesic effects and side effects (such as nausea-vomiting) were evaluated.

DETAILED DESCRIPTION:
The study was carried out with 60 ASA I-II class participants aged 20-60 years who underwent laparoscopic cholecystectomy at Van Yuzuncu Yıl University Faculty of Medicine. Preoperative evaluation was made before the operation, routine laboratory analyzes were taken, the participants were informed about the study, and their written consent was obtained. Participants were randomized into two groups.

* Group T (Adjuvant Tramadol): 40 mL of 0.250% bupivacaine + 1.5mg/kg and a maximum of 100 mg tramadol adjuvant
* Group D (Adjuvant Dexmedetomidine): 40 mL of 0.250% bupivacaine + 0.5 mcg/kg and a maximum of 50 mcg dexmedetomidine adjuvant Standard general anesthesia was applied. After intubation, bilateral subcostal TAP block was performed by the same anesthesiologist, demographic data were recorded. Intraoperative vital signs of the participants (pulse, non-invasive blood pressure and peripheral oxygen saturation measurement), additional opioid and muscle relaxant needs, and complications were recorded. Extubation was performed after standard decurarization with atropine and neostigmine. Postoperative side effects (nausea, vomiting, pruritus, shivering), postoperative additional analgesic need, and 0 hour (Modified aldrete score ≥9 time was accepted as 0 hour), 3rd hour and 6th hour Visual Analogue Scale (VAS) scores were evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years old
* Those who will undergo elective laparoscopic cholecystectomy surgery
* Those in ASA I-II physical status
* Those who gave consent to participate in the study

Exclusion Criteria:

* Those outside the age range of 20-60
* Those outside of ASA I-II physical status
* Serious heart, lung, liver disease
* Kidney failure
* Bleeding diathesis
* Those who develop complications during the procedure
* Those with fever, active infection
* Those who are allergic to the drugs to be used
* Those who refused to participate in the study
* Those with hypothermic and acid-base disorders
* Electrolyte disturbances such as hypokalemia, hypocalcemia
* Those taking antibiotics, anticonvulsants, antiarrhythmics, cholinesterase inhibitors
* Pregnant
* Those with bleeding
* BMI 30 and above

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
intraoperative non invasive blood pressure | 10 minutes
  non invasive blood pressure(systolic, diastolic and mean blood pressure)
intraoperative opioid consumption | 40 minutes
  The necessary opioid (mcg) addiction was noted
intraoperative muscle relaxant use | 40 minutes
  The necessary muscle relaxant (mg) addiction was noted
intraoperative heart rate | 5 minutes
  Heart rate was noted

SECONDARY OUTCOMES:
postoperative analgesic effects | 0., 3., 6. hour measurements were evaluated
  Visual analogue scale (VAS) scores were noted.pointed between 0-10. 0:No pain, 5-6-7:medium pain, 9-10:unbearable pain
Number of participants with postoperative side effects | 0., 3., 6. hour measurements were evaluated
  nausea, vomiting, chills. Patients with these effects were noted. Evaluated by the number of people

CONTACTS AND LOCATIONS:
Overall Officials: School of Medicine Department of Anesthesiology and Reanimation, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Korkutata Z, Tekeli AE, Kurt N. Intraoperative and Postoperative Effects of Dexmedetomidine and Tramadol Added as an Adjuvant to Bupivacaine in Transversus Abdominis Plane Block. J Clin Med. 2023 Nov 9;12(22):7001. doi: 10.3390/jcm12227001. PMID 38002616